CLINICAL TRIAL: NCT07093021
Title: Feasibility of Implementing the COLA-6 Case-Finding Tool to Identify Chronic Respiratory Disease in Primary Health Care in Brazil
Brief Title: Mitigating Chronic Respiratory Disease Through the Lens of Multimorbidity
Acronym: MARES2
Status: Not yet recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Universidade Federal de Sao Carlos (Other)
Responsible Party: Sponsor
Other Study IDs: 6981600 (UCL Worktribe); NIHR 303125 (Other Grant/Funding Number: UK NIHR (National Institute for Health and Care Research))
Record Dates: First submitted 2025-07-18; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Asthma; Preserved Ratio Impaired Spirometry
Keywords: case-finding; chronic obstructive pulmonary disease; asthma; multi-morbidity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aim to evaluate whether it is feasible for healthcare professionals to implement a case-finding tool to identify individuals at high risk for chronic respiratory diseases (CRDs) during routine care for non-communicable diseases (NCDs) in primary healthcare services in Brazil.

The investigators will complete a cross-sectional observational study involving 20 healthcare professionals (physicians, physiotherapists, community health agents, and nurses) from five primary healthcare services who will apply the COLA-6 tool during routine NCD care. A total sample of 1,000 patients is expected. Qualitative interviews will be conducted with healthcare professionals to explore barriers and facilitators to implementing COLA-6 in clinical practice.

DETAILED DESCRIPTION:
The investigators will assess the feasibility of healthcare professionals implementing the COLA-6 case-finding tool to identify individuals at high-risk of chronic respiratory diseases (CRDs) in primary health care (PHC) settings for non-communicable disease (NCD) care in Brazil. CRDs include asthma and chronic obstructive pulmonary disease (COPD). The COLA-6 ("COPD in Low- and Middle-Income Countries Assessment") is a validated and simple case-finding strategy designed to identify individuals at risk for CRDs in low- and middle-income country (LMIC) settings.

The study will be carried out in PHC services, including Basic Health Units (BHUs) and Family Health Units (FHUs), located in the municipalities of São Carlos and São Paulo, both in the state of São Paulo, Brazil.

The study will include two main participant groups:

(1) individuals with one or more NCDs who receive care from PHC services, and (2) healthcare professionals (HCPs) working in these settings.

HCPs will be recruited from BHUs and FHUs in São Carlos and São Paulo.

Eligible patients with NCDs will be identified by HCPs during routine appointments for NCDs (e.g., hypertension, diabetes, etc.). All participants will provide written informed consent.

The study comprises two phases:

Phase 1 - Implementation of COLA-6:

Application of the COLA-6 tool: After receiving prior training from the research team, HCPs at the BHUs and FHUs will identify potentially eligible individuals with NCDs who attend PHC services and will administer the COLA-6 tool as part of their routine care. Participants identified as being at high risk for CRDs based on the COLA-6 results will receive a leaflet with basic guidance on accessing diagnostic and treatment services for respiratory conditions.

Fidelity Monitoring: Selected administration of the COLA-6 tool by each HCP will be observed by the research team to ensure adherence to protocol.

Phase 2 - Evaluation of Implementation:

Upon completion of the 50 COLA-6 applications, HCPs will participate in qualitative interviews conducted by the research team to explore the barriers and facilitators to implementation in routine PHC settings.

Interviews will be audio-recorded, transcribed verbatim, and anonymized prior to analysis. The questions will address feasibility aspects such as the time required to complete the questionnaire, difficulties encountered, clarity of the questions, uncertainties during integration of the tool into the work routine, and patient receptiveness.

The research team will work in five BHU/FHUs, with five HCPs at each unit, each administering COLA-6 to fifty patients.

Patients identified as being at high risk for CRDs will be asked if they can be contacted for future research.

Descriptive statistics will be used to characterize patient and professional samples. Quantitative analysis of fidelity data will report categorical variables as frequencies (percentages). The qualitative analysis of the interviews will follow Braun and Clarke, which consists of six phases: 1) Familiarization with the data set; 2) Coding; 3) Generation of initial themes; 4) Development and review of themes; 5) Refinement, definition and naming of themes; and 6) Writing.

ELIGIBILITY:
Inclusion Criteria:

HCP: providing care to people with NCDs in PHC settings in Brazil. PATIENTS: attending for NCD care at a PHC setting in Brazil.

Exclusion Criteria:

HCP: not received training to deliver COLA-6.

PATIENTS:

* not provided informed consent
* clinically unstable in the past month
* current pregnancy
* active tuberculosis or being on treatment for tuberculosis
* cognitive impairment that would prevent understanding of the case-finding tool
* contra-indications to lung function testing.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. HCPs providing NCD care in PHC services in Brazil.
  2. Patients attending for NCD care in PHC services in Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Barriers and facilitators to implementing the COLA-6 case-finding tool. | At study completion: qualitative interviews will be completed after each HCP has completed 50 uses of COLA-6.
  Barriers and facilitators to implementing the COLA-6 case-finding tool, assessed at qualitative interviews.

CONTACTS AND LOCATIONS:
Overall Officials: John R Hurst, PhD FRCP, Principal Investigator — University College London Hospitals; Renata G Mendes, DFisio, Principal Investigator — Federal University of Sao Carlos (UFScar), Brasil
Locations (2):
- Brazil (2):
  - Multiple primary care sites, São Carlos, São Paulo
  - Multiple primary care sites, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No
We have no plans to share individual responses from qualitative interviews.